CLINICAL TRIAL: NCT05638321
Title: Minimally Invasive Micro Sclerostomy (MIMS®) Inferonasal Procedure - Performance Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanoculis Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MMS EEU-5
Record Dates: First submitted 2022-11-27; First posted 2022-12-06 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-01

CONDITIONS: This Study is Conducted Under Inclusion/ Exclusion Criteria

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Arm 1 (Experimental): Eyes of subjects with uncontrolled (IOP > 20 mmHg) open-angle glaucoma (OAG), where IOP is not controlled when using maximum tolerated glaucoma medications
  Interventions: Device: MIMS
- Treatment Arm 2 (Experimental): Eyes of subjects with uncontrolled (IOP > 20 mmHg) open-angle glaucoma (OAG), who failed prior filtering procedure or had uncontrolled IOP on tolerated glaucoma medications [Treatment Arm 2 and Treatment Arm 3].
  Interventions: Device: MIMS
- Treatment Arm 3 (Experimental): Two (2) inferonasal sclerostomies will be performed by the MIMS® system in the eyes of subjects who failed prior filtering procedure or had uncontrolled IOP on tolerated glaucoma medications (i.e., refractory glaucoma).
  Interventions: Device: MIMS

INTERVENTIONS:
Device: MIMS — sterile surgical device made of stainless steel and plastic, which is coupled to a rotating system. The surgical device consists of stainless steel micro trephine, covered by a small needle and rotating mechanism behind it. Mechanical rotation of the surgical device is achieved by the rotating system which is comprised of a 1) Controller which dictates the activation pulse duration and RPM, 2) a Motor, and 3) Footswitch.

SUMMARY:
Minimally Invasive Micro Sclerostomy (MIMS®) device is intended for the reduction of elevated Intraocular Pressure (IOP).

MIMS® is a powered surgical device, designed to create a drainage channel of 100 microns diameter at the sclera-corneal junction and extending from the anterior chamber to the interface between the sclera and the conjunctiva (subconjunctival space), at the inferonasal quadrant of the eye (i.e., inferonasal sclerostomy).

The drainage channel is created by a sterile surgical device made of stainless steel and plastic, which is coupled to a rotating system. The surgical device consists of stainless steel micro trephine, covered by a small needle and rotating mechanism behind it. Mechanical rotation of the surgical device is achieved by the rotating system which is comprised of a 1) Controller which dictates the activation pulse duration and RPM, 2) a Motor, and 3) Footswitch.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years to ≤ 85 years old
2. Unsatisfactory IOP level, i.e., IOP ≥21 mmHg, at the screening visit in the study eye
3. Manifest open angle glaucoma (OAG) with typical disc or visual field changes and open iridocorneal angle in the study eye (in accordance with European Glaucoma Society (EGS) criteria 1)
4. Optic nerve appearance characteristic of glaucoma in the study eye
5. Shaffer grade ≥ III in all four angle quadrants in the study eye
6. Subject is treated with 0 to 5 hypotensive medications in the study eye
7. Subject is able and willing to attend all scheduled follow-up exams
8. Subject understands and signs the informed consent

   In addition, subjects meeting the following criterion will be considered for enrolment into Treatment Arm 2 or Treatment Arm 3 of the trial:
9. Subject with refractory glaucoma, defined as prior failure of filtering procedure and/or uncontrolled IOP on maximally tolerated medical therapy (i.e., ≥ 4 classes of topical IOP-lowering medications, or fewer in the case of tolerability or efficacy issues) . Specifically, subjects who:

   * Failed one or more incisional intraocular glaucoma surgeries (e.g., glaucoma filtering surgery);
   * Have neovascular glaucoma;
   * Have any other condition (e.g., conjunctival scarring, uveitis) in which a conventional incisional glaucoma surgery like trabeculectomy would be more likely to fail than for an eye with uncomplicated primary open angle glaucoma

Exclusion Criteria:

- Exclusion Criteria

Subjects presenting 1 or more of the following criteria will not be enrolled in any of the treatment arms of the trial:

1. Ocular conditions with a poorer prognosis in the fellow eye than in the study eye
2. Closed angle forms of glaucoma in either eye unless scheduled for cataract surgery immediately prior to the Minimally Invasive Nasal Trabeculostomy System procedure or the study eye is pseudophakic with posterior chamber intraocular lens (PCIOL)
3. Congenital or developmental glaucoma in either eye
4. Fixation threatening visual-field defects or IOP ≥40 mmHg in the study eye
5. Other secondary glaucoma (such as neovascular, uveitic, lens-induced, trauma-induced, or glaucoma associated with increased episcleral venous pressure) in the study eye
6. Peripheral anterior synechiae (PAS), rubeosis or other angle abnormalities in the study eye
7. Subject has history of penetrating keratoplasty (PKP)
8. Any ocular disease or history in study eye such as severe dry eye, active proliferative retinopathy, ICE syndrome, epithelial or fibrous down growth, and ocular pathology that may interfere with accurate IOP measurements
9. Prior surgery for an ab-interno or ab-externo device implanted in or through the Schlemm's canal in the study eye
10. Best-corrected visual acuity worse than 20/40 (Snellen equivalent) in the fellow eye
11. History of idiopathic or autoimmune uveitis in either eye
12. Severe trauma in study eye
13. Active iris neovascularization, previous cyclodestructive procedure, prior scleral buckling procedure, presence of silicone oil, need for glaucoma surgery combined with other ocular procedures or anticipated need for additional ocular surgery in study eye within 12 month period
14. Vitreous present in anterior chamber, prior vitrectomy or vitreous hemorrhage in study eye
15. Aphakia
16. Prior vitreoretinal surgery in study eye
17. Clinically significant ocular inflammation or infection within 90 days prior to screening
18. Unable to discontinue use of blood thinners in accordance with surgeon's standard preoperative instructions
19. Uncontrolled systemic disease that in the opinion of the investigator would put the subject's health at risk and/or prevent the subject from completing all study visits
20. Current participation or participation in another investigational drug or device clinical trial within the last 30 days before screening visit
21. Pregnant or lactating women

    Additionally, subjects presenting 1 or more of the following criteria will not be enrolled in Treatment Arm 1 of the trial:
22. Prior glaucoma filtering surgery, such as trabeculectomy, in the study eye
23. Prior cilioablative procedure in the study eye

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a 20% or greater reduction in IOP from baseline on the same or fewer number of medications at 24-week visit | 24 weeks
  • Proportion of subjects achieving a 20% or greater reduction in IOP from baseline on the same or fewer number of medications. Subjects who will undergo reoperation for glaucoma prior to the 24 weeks visit will be considered failures in the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- S.V.Malayan'S Eye Center, Yerevan, Armenia